CLINICAL TRIAL: NCT05877976
Title: Impact of Visual Arts Immersion on Cultural Competency and Self-reflection Among Nurses Working in an Academic Health System
Brief Title: Impact of Visual Arts Immersion
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Collaborators: National Library of Medicine (NLM) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 23-00530
Record Dates: First submitted 2023-05-18; First posted 2023-05-26 (Actual); Results first posted 2025-01-22 (Actual); Last update posted 2025-01-22 (Actual); Status verified 2024-12

CONDITIONS: Cultural Competency; Personal Reflection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Registered Nurses (Experimental): Participants will receive an intervention of museum educator-led workshops that introduce nurses to arts appreciation skills to improve their practice and overall wellbeing.
  Interventions: Behavioral: Visual Arts Immersion

INTERVENTIONS:
Behavioral: Visual Arts Immersion — Museum educators from The Metropolitan Museum of Art (MET) will provide a curriculum including an art immersion program that will select specific works/art in the museum as well as virtually that will help to stimulate self-reflection and prompt connection to their nursing practice. Participants will be asked to sign up for 2 art immersion classes. The first class will be an in-person class at The MET and the second class will be virtual via WebEx. Each class will last 60 minutes.

SUMMARY:
The purpose of this study is to enhance engagement, coping and self-reflection by attuning nurses to creative and observational skills drawn from a visual arts pedagogical framework. To fulfill this goal, the investigators will cultivate an existing relationship between NYU Langone Health (NYULH) Nursing, the NYU Health Sciences Library, and museum educators at The Met to design and deliver an intervention of museum educator-led workshops that introduce nurses to arts appreciation skills to improve their practice and overall wellbeing. Participants will be asked to complete two surveys, pre- and post-intervention, Cultural Awareness Scale (CAS), which measures cultural awareness, sensitivity, knowledge and skills, and the Interpersonal Reactivity Index (IRI), which measures four separate aspects of empathy and its relationships with measures of social functioning, self-esteem, emotionality, and sensitivity to others. We will also solicit qualitative feedback via REDCap survey at the end of the intervention to gain insight into nurse's experiences of the art immersion program.

ELIGIBILITY:
Inclusion Criteria:

1. A Registered Nurse at NYULH
2. Willing to provide an email address or cell phone number of choice
3. Willing to attend one workshop in person at The MET and one virtually via WebEx
4. Willing and able to provide consent
5. Age 18 years of age or older

Exclusion Criteria:

1. Not a Registered Nurse at NYULH
2. Not willing to provide an email address or cell phone number of choice
3. Not willing to attend one workshop in person at The MET and one virtually via WebEx

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2023-06-15 (Actual); Primary Completion 2024-03-21 (Actual); Study Completion 2024-03-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lita Anglin, Principal Investigator — NYU Langone Health
Locations (1):
- NYU Langone Health, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No
This study is only open to NYU Langone Health Employees.

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Registered Nurses
Started | 41
Completed | 10
Not Completed | 31
Not completed — Lost to Follow-up | 31

BASELINE CHARACTERISTICS:
Arm/Group | Registered Nurses
Number analyzed (Participants) | 10
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.2 (16.75)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 10
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 7
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 10

OUTCOME MEASURES:

1. Primary Outcome: Change in Cultural Awareness Scale (CAS) Score From Baseline to Month 6
Description: 36-item questionnaire assessing cultural awareness, sensitivity, knowledge and skills. Each item is rated on a 7-point scale (ranging from "strongly disagree" to "strongly agree"). The total score ranges from 0-252. Lower scores indicate less cultural awareness, and higher scores indicate greater awareness.
Time Frame: Baseline, Month 6
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Registered Nurses
Number analyzed (Participants) | 10
score on a scale | 11.90 [-1.32 to 25.12]

2. Primary Outcome: Change in Clinical Interpersonal Reactivity Index (CIRI) Score From Baseline to Month 6
Description: 27-item questionnaire evaluating empathy as a reaction in interpersonal relationships at the bedside. Items are ranked on a scale from 0-4, where 0 = does not describe me well; and 4 = describes me very well. The total score ranges from 0 to 108; higher scores indicate greater empathy.
Time Frame: Baseline, Month 6
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Registered Nurses
Number analyzed (Participants) | 10
score on a scale | 4.7 [0.10 to 9.30]

ADVERSE EVENTS:
Time Frame: Month 6
Description: At each contact with the subject, the investigator must seek information on adverse events by specific questioning and, as appropriate, by examination.
Arm/Group | Registered Nurses
All-Cause Mortality (participants affected / at risk) | 0/41
Serious Adverse Events (participants affected / at risk) | 0/41
Other Adverse Events (participants affected / at risk) | 0/41

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-01-16): https://cdn.clinicaltrials.gov/large-docs/76/NCT05877976/Prot_SAP_001.pdf
  • Informed Consent Form (2023-06-19): https://cdn.clinicaltrials.gov/large-docs/76/NCT05877976/ICF_000.pdf